CLINICAL TRIAL: NCT04041713
Title: A Pilot Study of an Antioxidant Cocktail vs. Placebo in the Treatment of Children and Adolescents With Rett Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Ontario Brain Institute (Other); Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RETT-08-2018
Record Dates: First submitted 2019-06-27; First posted 2019-08-01 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Rett Syndrome
Keywords: Rett Syndrome; Rett; RTT
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Intervention Model Description: This is an 18-week pilot, single site, randomized,double blind, placebo-controlled cross-over trial of Rett-T vs. placebo. Periods I and II of the randomized study are 8 weeks long with a 2 week washout period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rett T (Active Comparator): Rett T is a powder for oral suspension. Dosage is dependent on weight. For participants weighing <30 kg, a 4 g dose (i.e., one 4 g sachet) is intended to be administered orally once a day after dissolving in approximately 125 mL of water. For participants weighing ≥30 kg, a 8 g dose (i.e., two 4 g sachets) is intended to be administered orally once a day after dissolving in approximately 250 mL of water.
  Interventions: Drug: Rett-T
- Placebo (Placebo Comparator): Placebo is a powder for oral suspension. Dosage is dependent on weight. For participants weighing <30 kg, a 4 g dose (i.e., one 4 g sachet) is intended to be administered orally once a day after dissolving in approximately 125 mL of water. For participants weighing ≥30 kg, a 8 g dose (i.e., two 4 g sachets) is intended to be administered orally once a day after dissolving in approximately 250 mL of water.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rett-T — antioxidant cocktail
  Arms: Rett T
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will examine the potential efficacy and safety of Rett-T for core motor deficits of Rett syndrome, and will explore biological markers of safety and treatment response.

DETAILED DESCRIPTION:
There are currently no available medicines shown to be effective for Rett syndrome. Numerous studies implicate mitochondrial dysfunction and oxidative stresses in the pathophysiology of Rett syndrome. Mitochondrial dysfunction has been reported in Rett patients, Rett mouse models and MECP2-deficient cells.

Collaborators have tested a combination of specific antioxidants known to enhance mitochondrial function in a cell and mouse model of Rett syndrome. The formulation normalized mitochondrial membrane potential in MECP2 neurons, and MECP2-deficient mice displayed improved exploratory, locomotor and social behavior compared to MECP2-deficient mice. These results support testing anti-oxidative strategies for benefit in individuals with Rett syndrome.In this study, the formulation has been adjusted and optimized based on current guidelines for human use, with the goal of translating a potential new treatment from the animal model to use in humans. Results of this study could lead to the first approved medication treatment for the disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Female outpatients 2-21 years of age inclusive.
2. Diagnosis of Rett syndrome.
3. At least partially ambulatory (may need assistive device to take a step).
4. If already receiving stable interventions must meet the following criteria:

   * If already receiving stable concomitant medications or nutraceuticals affecting behaviour, must be on a stable dose during the preceding 1 month prior to Screening (with the exception of fluoxetine, where a period of 6 weeks is needed), and will not electively initiate new or modify ongoing medications for study duration.
5. Have normal laboratory test results at Screening/Baseline. If abnormal, the finding(s) must be deemed clinically insignificant by the Investigator.
6. Ability to complete assessments, fluency in English (parent/legal guardian; participant, if verbal).
7. Ability to obtain assent (if developmentally appropriate), as well as written informed consent from their parent(s)/legal guardian(s).

Exclusion Criteria:

1. Pregnant females; sexually active females on inadequate birth control (extremely unlikely in this population).
2. Have another serious medical condition that, based on Investigator judgment, might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. Have evidence or history of malignancy or any significant hematological, endocrine, cardiovascular (including any rhythm disorder), respiratory, renal, hepatic, or gastrointestinal disease, not including mild common pediatric diseases in these areas that are stable (e.g. mild asthma, constipation, etc.).
3. Have hypersensitivity to any components of Rett-T.
4. Have one or more of the following: HIV, HBV, HCV, hemophilia (bleeding problems, recent nose and brain injuries), drug abuse, immunity disorder, major depressive episode or psychosis.
5. Unable to tolerate venipuncture procedures for blood sampling.
6. Receiving concomitant medications/nutraceuticals that include any of the components of Rett-T.
7. Actively enrolled in another intervention study.

Ages: 2 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Rett Syndrome Natural History Motor Behavior Assessment (MBA) | 18 weeks total: 8 weeks on Rett-T, 8 weeks on placebo, 2 week washout in interim
  To examine the effect of Rett-T vs. placebo on measures of motor function. The Rett Syndrome MBA consists of 37 items grouped into three subscales (Behavioral/Social Assessment, Orofacial Respiratory Assessment, and Motor Assessment/Physical Signs). Items are captured on a 0-4 point Likert scale. Total and subscale scores are calculated (subscales are summed for a total score). The scale range for Total score is 0-136; for Behavioral/Social subscale, 0-60; for Orofacial/Respiratory subscale, 0-28; for Motor Assesment/Physical Signs, 0-48. For both total and subscale scores, higher values represent a worse outcome.

SECONDARY OUTCOMES:
Rett Syndrome Gross Motor Scale (RSGMS) | 18 weeks total: 8 weeks on Rett-T, 8 weeks on placebo, 2 week washout in interim
  To examine the effect of Rett-T vs. placebo on measures of motor function. The RSGMS consists of 15 gross motor items grouped into three subscales (Sitting, Standing and Walking, and Challenge). Items are captured on a 0-3 Likert Scale rating regarding level of assistance needed (0=maximal, 3 = none). Total and subscale scores are calculated (subscales are summed for a total score). The scale range for Total score is 0-45; for Sitting, 0-9; for Walking, 0-27; for Challenge, 0-9. For both total and subscale scores, higher values represent a better outcome.
Safety Monitoring Uniform Report Form (SMURF) | 18 weeks total: 8 weeks on Rett-T, 8 weeks on placebo, 2 week washout in interim
  To examine the safety and tolerability of Rett- T in children and youth with Rett syndrome; To explore the effect Rett-T vs. placebo on maladaptive behaviors, anxiety, sleep, seizure
Clinical Global Impressions - Improvement Scale - Global (CGI-I) | 18 weeks total: 8 weeks on Rett-T, 8 weeks on placebo, 2 week washout in interim
  To explore the effect of Rett-T vs. placebo on global improvement. The CGI-I measures global clinical improvement in response to treatment. A single score is assigned on a 1-7 Likert scale, with 1= very much improved-7=very much worse. Higher values represent a worse outcome.
The Top 3 Causes for Concern | 18 weeks total: 8 weeks on Rett-T, 8 weeks on placebo, 2 week washout in interim
  To explore the effect Rett-T vs. placebo on maladaptive behaviors, anxiety, sleep, seizure frequency, and global improvement. Respondents are instructed to choose their top three concerns for the participant, and indicate Concern Number #1, 2 and 3 on the form. Respondents are next instructed to place a vertical mark along a visual analogue scale (a 10 centimetre horizontal line in which the leftmost point on the scale indicates the concern is completely absent, and the rightmost point on the scale indicates that the concern is very severe). For each concern, a measurement is taken from the leftmost point of the scale to the vertical mark, and the measurement in centimetres acts as the score. Higher scores represent a worse outcome.
The Rett Syndrome Behaviour Questionnaire (RSBQ) | 18 weeks total: 8 weeks on Rett-T, 8 weeks on placebo, 2 week washout in interim
  To explore the effect of Rett-T vs. placebo on maladaptive behaviors, anxiety, sleep, seizure frequency, and global improvement. The measure consists of 45 items which are grouped into 8 subscales (General Mood, Breathing Problems, Body Rocking and Expressionless Face, Hand Behaviors, Repetitive Face Movements, Night-time Behaviors, Fear/Anxiety, and Walking/Standing). Items are measured on a 0-2 Likert scale.Total and subscale scores are calculated (subscales are summed for a total score). The scale range for total score is 0-90; for General Mood, 0-16; for Breathing Problems, 0-10; for Body Rocking and Expressionless Face, 0-12; for Hand Behaviours, 0-12; for Repetitive Face Movements, 0-8; for Nighttime Behaviours, 0-6; for Fear/Anxiety; 0-8; for Walking/Standing, 0-4. Seven items are not included in the subscale scores but are included in the total score sum. For both total and subscale scores, higher values represent a worse outcome.
Anxiety, Depression, and Mood Scale (ADAMS) | 18 weeks total: 8 weeks on Rett-T, 8 weeks on placebo, 2 week washout in interim
  To explore the effect of Rett-T vs. placebo on anxiety. The ADAMS consists of 28 items grouped into five subscales (Manic/Hyperactive Behavior, Depressed Mood, Social Avoidance, General Anxiety, and Obsessive Behavior). Items are scored on a 0-3 Likert scale that combines frequency and severity ratings (where 0=behavior has not occurred or is not a problem, 3=behavior occurs a lot or is a severe problem). Each subscale score is calculated separately; the scale range for Manic/Hyperactive Behavior is 3-15; for Depressed Mood, 7-21; for Social Avoidance, 7-21; for General Anxiety, 7-21; for Obsessive Behavior, 3-9. For each subscale score, higher values represent a worse outcome.
Children's Sleep Habits Questionnaire (CSHQ) | 18 weeks total: 8 weeks on Rett-T, 8 weeks on placebo, 2 week washout in interim
  To explore the effect of Rett-T vs. placebo on sleep. The CSHQ is a tool designed to screen for the most common sleep problems in children. The CSHQ consists of 35 items for scoring and extra unscored items intended to provide administrators with other potentially useful information about respondents. The instrument evaluates sleep based on behavior within eight different subscales (Bedtime Resistance, Sleep-Onset Delay, Sleep Duration, Sleep Anxiety, Night Wakings, Parasomnias, Sleep-Disordered Breathing, and Daytime Sleepiness).Total and subscale scores are calculated (33 items are summed for a total score). The scale range for Total score is 33-99; for Bedtime Resistance subscale, 6-18; for Sleep Onset/Delay, 1-3; for Sleep Duration, 3-9; for Sleep Anxiety, 4-12; For Night Wakings, 3-9; for Parasomnias, 7-21; for Sleep-Disordered Breathing, 3-9; for Daytime Sleepiness, 8-24. For both total and subscale scores, higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, MD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No